CLINICAL TRIAL: NCT01898078
Title: An Open-Label, Phase 1, Two-Way, Cross-Over Study of the Effect of the Food on the Pharmacokinetics of MLN8237 (Alisertib) in Patients With Advanced Solid Tumors or Lymphomas
Brief Title: Food Effect Study of Alisertib (MLN8237) in Participants With Advanced Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C14017
Record Dates: First submitted 2013-07-01; First posted 2013-07-12 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-03

CONDITIONS: Advanced Solid Tumors; Lymphoma
Keywords: MLN8237; Alisertib; Food effects
MeSH Terms: conditions — Lymphoma | interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alisertib 50 mg Fed + Fasted (Experimental): Alisertib 50 mg, enteric-coated tablets (ECT), orally, in fed state, once on Day 1, followed by alisertib 50 mg, ECT, orally, twice daily (BID) on Days 4 through 10, followed by a 14-day rest period in Cycle 1 (24-day cycles), followed by alisertib 50 mg, ECT, orally, in fasted state, once on Day 1, followed by alisertib 50 mg, ECT, orally, BID on Days 4 through 10, followed by a 14-day rest period in Cycle 2, followed by alisertib 50 mg, ECT, orally, BID on Days 1-7, followed by a 14-day rest period in Cycle 3 and onwards (21-day cycles) until disease progression, occurrence of an unacceptable alisertib-related toxicity.
  Interventions: Drug: Alisertib
- Alisertib 50 mg Fasted + Fed (Experimental): Alisertib 50 mg, ECT, orally, in fasted state, once on Day 1, followed by alisertib 50 mg, ECT, orally, BID on Days 4 through 10, followed by a 14-day rest period in Cycle 1 (24-day cycles), followed by alisertib 50 mg, ECT, orally, in fed state, once on Day 1, followed by alisertib 50 mg, ECT, orally, BID on Days 4 through 10, followed by a 14-day rest period in Cycle 2, followed by alisertib 50 mg, ECT, orally, BID on Days 1-7, followed by a 14-day rest period in Cycle 3 and onwards (21-day cycles) until disease progression, occurrence of an unacceptable alisertib-related toxicity.
  Interventions: Drug: Alisertib

INTERVENTIONS:
Drug: Alisertib — Alisertib ECT
  Other Names: MLN8237

SUMMARY:
The purpose of this study is to evaluate the effect of food on the single-dose pharmacokinetics (PK) of alisertib administered as an enteric-coated tablet (ECT) formulation in participants with advanced solid tumors or lymphomas.

DETAILED DESCRIPTION:
The drug being tested in this study is called alisertib. Alisertib is being tested in adult participants with advanced solid tumors or lymphomas.

The study enrolled 26 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Alisertib 50 mg Fed + Fasted
* Alisertib 50 mg Fasted + Fed

All participants will be asked to take one alisertib tablet (ECT), orally, with or without a standard high-fat breakfast Cycle 1, Day 1, with the respective alternate food intake condition (fasted to fed or fed to fasted) on Cycle 2, Day 1, each followed by 14-day rest period. Participants will take alisertib, ECT, orally BID on Days 4 to 10 of Cycles 1 and 2, each followed by 14-day rest period. From Cycle 3 onwards participants will continue taking alisertib 50 mg, ECT, orally, BID on Days 1-7, followed by a 14-day rest period in 21-day cycles until disease progression, occurrence of an unacceptable alisertib-related toxicity.

This multi-center trial conducted at 3 sites in the United States. Participants will make multiple visits to the clinic and plus a final visit after 30 days of receiving their last dose of drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Histologically or cytologically confirmed advanced tumors or lymphomas for which standard curative or life-prolonging treatment does not exist, or is no longer effective or tolerable
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Participant must meet protocol-specified laboratory values
* Suitable venous access
* Female participants who are postmenopausal for at least 1 year OR are surgically sterile OR if of childbearing potential, agree to practice 2 effective methods of contraception at the same time or agree to practice true abstinence
* Male participants who agree to practice effective barrier contraception during the entire study and through 4 months after the last dose of study drug OR agree to practice true abstinence

Exclusion Criteria:

* Prior or current investigational therapies within 4 weeks before the first dose of alisertib
* Female participants who are lactating or pregnant
* Participant requiring treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine, or phenobarbital, or rifampin, rifabutin, rifapentine, or St. John's wort within 14 days before the first dose of alisertib and during the study
* Medical conditions requiring daily, chronic, or regular use of proton pump inhibitors (PPIs) within 7 days preceding the first dose of alisertib, or histamine (H2)-receptor antagonists
* Participant requiring systemic anticoagulation
* Ongoing nausea or vomiting that is Grade 2 or worse in intensity
* Known gastrointestinal (GI) disease or GI procedures that could interfere with the oral absorption, excretion, or tolerance of alisertib
* History of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness such as severe chronic obstructive pulmonary disease
* Known or suspected human immunodeficiency virus (HIV) positive or hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection
* Participant who are lactose-intolerant or are unwilling/unable to consume the protocol specified standardized high-fat breakfast

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-07-16 (Actual); Primary Completion 2014-03-05 (Actual); Study Completion 2017-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - The Bronx, New York
  - Nashville, Tennessee
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in the United States from 16 July 2013 to 24 January 2017. Data cut-off for the primary analysis was 05 March 2014.
Pre-assignment Details: Participants with a diagnosis of advanced solid tumors or lymphomas were enrolled to crossover fashion to receive alisertib 50 mg enteric-coated tablet (ECT), orally in fasted or fed state in Cycles 1 and 2.
Period: Overall Study
Arm/Group | Alisertib 50 mg Fed + Fasted | Alisertib 50 mg Fasted + Fed
Started | 13 | 13
Completed | 7 (Completed treatment) | 5 (Completed treatment)
Not Completed | 6 | 8
Not completed — Progressive Disease | 1 | 5
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Symptomatic Deterioration | 2 | 0
Not completed — Reason not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alisertib 50 mg Fed + Fasted | Alisertib 50 mg Fasted + Fed | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (10.15) | 61.7 (12.64) | 60.7 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 7 | 6 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 8 | 9 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 13 | 23
  Black or African American | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 13 | 26
Height [Mean (Standard Deviation); unit: cm] | 166.9 (14.34) | 165.3 (11.32) | 166.1 (12.68)
Weight [Mean (Standard Deviation); unit: kg] | 73.59 (15.484) | 78.37 (20.183) | 75.98 (17.792)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration of Alisertib
Time Frame: Cycles 1 and 2, Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: Pharmacokinetic (PK) population included participants with sufficient dosing data and PK concentration-time data to reliably estimate the PK parameters.
Measure: Mean (Standard Deviation); unit: nM
Groups:
- Alisertib 50 mg Fed: Alisertib 50 mg, ECT, orally, in fed state, once on Day 1 in Cycles 1 and 2.
- Alisertib 50 mg Fasted: Alisertib 50 mg, ECT, orally, in fasted state, once on Day 1 in Cycles 1 and 2.
Arm/Group | Alisertib 50 mg Fed | Alisertib 50 mg Fasted
Number analyzed (Participants) | 22 | 22
nM | 1338.6 (487.25) | 1354.5 (432.17)
Statistical Analysis 1: Comparison: Alisertib 50 mg Fed vs Alisertib 50 mg Fasted; The confidence intervals are calculated for the difference in the LS means of the ln-transformed Cmax plain values (difference = Fed/Fasted). Antilogs of the confidence limits for the difference are taken to construct the confidence intervals for the ratio of the geometric means; Test type: Superiority or Other; Least Squares Mean Ratio = 0.97, 90% CI 2-sided [0.85 to 1.12] — Estimates for each PK parameter were obtained using a mixed effects model of log (PK parameter) with fixed terms for the treatment effect, sequence effect, period effect and random terms for participants within sequence

2. Primary Outcome: AUC(Last): Area Under the Plasma Concentration Curve From Time 0 to the Time of the Last Quantifiable Concentration of Alisertib
Time Frame: Cycles 1 and 2, Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: PK population included participants with sufficient dosing data and PK concentration-time data to reliably estimate the PK parameters.
Measure: Mean (Standard Deviation); unit: hr*nM
Arm/Group | Alisertib 50 mg Fed | Alisertib 50 mg Fasted
Number analyzed (Participants) | 22 | 22
hr*nM | 24645.5 (12467.39) | 20797.7 (8847.69)
Statistical Analysis 1: Comparison: Alisertib 50 mg Fed vs Alisertib 50 mg Fasted; The confidence intervals are calculated for the difference in the LS means of the ln-transformed AUC(last) plain values (difference = Fed/Fasted). Antilogs of the confidence limits for the difference are taken to construct the confidence intervals for the ratio of the geometric mean; Test type: Superiority or Other; Least Square Mean Ratio = 1.16, 90% CI 2-sided [1.01 to 1.34] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration Curve From Time 0 to Infinity of Alisertib
Time Frame: Cycles 1 and 2, Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: PK population included participants with sufficient dosing data and PK concentration-time data to reliably estimate the PK parameters. Here, number of participants analysed are the participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hr*nM
Arm/Group | Alisertib 50 mg Fed | Alisertib 50 mg Fasted
Number analyzed (Participants) | 16 | 14
hr*nM | 24537.5 (9882.10) | 22771.4 (10206.21)
Statistical Analysis 1: Comparison: Alisertib 50 mg Fed vs Alisertib 50 mg Fasted; The confidence intervals are calculated for the difference in the LS means of the ln-transformed AUC∞ plain values (difference = Fed/Fasted). Antilogs of the confidence limits for the difference are taken to construct the confidence intervals for the ratio of the geometric mean; Test type: Superiority or Other; Least Square Mean Ratio = 1.15, 90% CI 2-sided [0.96 to 1.39] — Estimates for each PK parameter were obtained using a mixed effects model of log(PK parameter) with fixed terms for the treatment effect, sequence effect, period effect and random terms for participants within sequence

4. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study were reported as adverse events.
  A SAE is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: From first dose through 30 days after the last dose of study drug (up to 225 days)
Population: Safety population included all enrolled participants who received at least one dose of study drug. According to the protocol analysis planned, data for the safety and tolerability was collected as per the treatment sequence received in the study, irrespective of the fed or fasted condition.
Measure: Count of Participants; unit: Participants
Arm/Group | Alisertib 50 mg Fed + Fasted | Alisertib 50 mg Fasted + Fed
Number analyzed (Participants) | 13 | 13
Participants
  AEs | 13 | 13
  SAEs | 7 | 7

5. Secondary Outcome: Number of Participants With Clinically Significant Change in Laboratory Parameters Reported as AEs
Description: The number of participants with any clinical significant change in safety laboratory values collected throughout the study.
Time Frame: From first dose through 30 days after the last dose of study drug (up to 225 days)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Alisertib 50 mg Fed + Fasted | Alisertib 50 mg Fasted + Fed
Number analyzed (Participants) | 13 | 13
Participants
  Neutropenia | 10 | 8
  Anaemia | 5 | 3
  Leukopenia | 5 | 2
  Thrombocytopenia | 1 | 2
  Hypokalaemia | 0 | 3
  Hyperbilirubinaemia | 1 | 1
  Neutrophil count decreased | 1 | 1
  Lymphopenia | 0 | 1
  Hyperkalaemia | 1 | 0
  Hypomagnesaemia | 0 | 1
  Aspartate aminotransferase increased | 0 | 1
  Blood bilirubin increased | 1 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Change in Vital Sign Reported as AEs
Description: The number of participants with any clinical significant change in vital signs (sitting diastolic and systolic blood pressure, heart rate, and temperature) were collected throughout the study.
Time Frame: From first dose through 30 days after the last dose of study drug (up to 225 days)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Alisertib 50 mg Fed + Fasted | Alisertib 50 mg Fasted + Fed
Number analyzed (Participants) | 13 | 13
Participants
  Hypertension | 0 | 1
  Hypotension | 0 | 1
  Tachycardia | 0 | 1

ADVERSE EVENTS:
Time Frame: From first dose through 30 days after the last dose of study drug (up to 225 days)
Description: According to the protocol analysis planned, data for the safety and tolerability was collected as per the treatment sequence received in the study, irrespective of the fed or fasted condition.
Arm/Group | Alisertib 50 mg Fed + Fasted | Alisertib 50 mg Fasted + Fed
All-Cause Mortality (participants affected / at risk) | 0/13 | 1/13
Serious Adverse Events (participants affected / at risk) | 7/13 | 7/13
Other Adverse Events (participants affected / at risk) | 13/13 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib 50 mg Fed + Fasted (N=13) | Alisertib 50 mg Fasted + Fed (N=13)
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 — One treatment emergent death occurred during treatment with Alisertib 50 mg Fasted + Fed arm and is not related to the study drug.
Cellulitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib 50 mg Fed + Fasted (N=13) | Alisertib 50 mg Fasted + Fed (N=13)
Tachycardia (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 2 | 0
Eyelid cyst (Eye disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Micturition urgency (Renal and urinary disorders) | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Genital herpes (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Vaginitis bacterial (Infections and infestations) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 11 | 8
Anaemia (Blood and lymphatic system disorders) | 6 | 4
Leukopenia (Blood and lymphatic system disorders) | 5 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 1 | 2
Somnolence (Nervous system disorders) | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Fatigue (General disorders) | 8 | 3
Pyrexia (General disorders) | 1 | 5
Asthenia (General disorders) | 1 | 3
Oedema peripheral (General disorders) | 1 | 2
Chills (General disorders) | 1 | 1
Local swelling (General disorders) | 2 | 0
Catheter site erythema (General disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 1 | 0
Catheter site pain (General disorders) | 1 | 0
Infusion site vesicles (General disorders) | 1 | 0
Localised oedema (General disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoe (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 8
Vomiting (Gastrointestinal disorders) | 3 | 7
Diarrhoea (Gastrointestinal disorders) | 5 | 4
Nausea (Gastrointestinal disorders) | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 7
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculovesicular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.